CLINICAL TRIAL: NCT02016157
Title: Moxifloxacin In Situ Gel as an Adjunct in the Treatment of Periodontal Pocket: A Randomized Clinical Trial.
Brief Title: Moxifloxacin in Situ Gel to Treat Periodontal Pocket.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sri Hasanamba Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr. Shaurya Manjunath, Shaurya Manjunath, Post graduate Student, Department of Periodontology, Sri Hasanamba Dental College and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shaurya Manjunath
Record Dates: First submitted 2013-11-06; First posted 2013-12-19 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Chronic Generalized Periodontitis
Keywords: Moxifloxacin; Chlorhexidine; In situ gel; Chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Moxifloxacin, Chronic periodontitis (Experimental): 50 micrograms Moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Moxifloxacin — TO ASSESS THE EFFICACY OF MOXIFLOXACIN IN SITU GEL IN THE TREATMENT OF PERIODONTAL POCKET.
  Other Names: Avelox

SUMMARY:
In this Randomized clinical trial locally delivered moxifloxacin in situ gel was evaluated as an adjunct to scaling and root planing for efficacy in the treatment of chronic periodontitis and for short-term effects on the periodontal microflora.

DETAILED DESCRIPTION:
Moxifloxacin exerts excellent antibacterial activity against a wide range of putative periodontal pathogens, including Porphyromonas gingivalis, Tannerella forsythia, Prevotella species, Fusobacterium nucleatum, Actinomyces species, Peptostreptococcus species, Campylobacter rectus, and Actinobacillus actinomycetemcomitans. Moxifloxacin penetrates well into soft tissues and is effective against intracellular periodontal pathogens when used in the treatment of periodontitis as an adjunct to scaling and root planning (SRP). Systemic administration of moxifloxacin has provided superior outcomes compared with SRP in conjunction with systemic administration of doxycycline, or SRP alone. We hypothesized similar benefits with local drug delivery of Moxifloxacin in the treatment of chronic periodontitis. To the best of our knowledge, there is no published literature on in situ gel using moxifloxacin employing gellan gum as the vehicle, for direct placement in the periodontal pocket for the treatment of chronic periodontitis.

Among various drug delivery systems for treating periodontitis, gel formulations have some advantages. Despite a relatively faster release of the drug, gels can be more easily prepared and administered. Moreover, they possess a higher bio compatibility and bio adhesivity, by allowing adhesion to the mucosa in the dental pocket and by decreasing the risk of dilution of the material by saliva.

Keeping the above facts in mind, the goals of this study were to (1) evaluate in situ gel as a vehicle in a local drug delivery system, (2) evaluate the efficacy of moxifloxacin for local drug delivery, (3) evaluate the efficacy of gellan gum for in situ gelation of moxifloxacin, and (4) evaluate and compare the clinical and microbiological parameters of moxifloxacin with those of the gold standard, chlorhexidine di gluconate.

ELIGIBILITY:
Inclusion Criteria:

* patients with good systemic health
* Patients with Chronic periodontitis with sites with probing pocket depth (PPD) of ≥ 5 mm
* a minimum of 12 natural teeth with radiographic evidence of bone loss
* willingness to comply with the study protocol.

Exclusion Criteria:

* Patients with a history of drug allergy to quinolones or those who were taking medication that might interact with moxifloxacin
* Patients with history of antibiotic coverage in the 6 months preceding the study
* Pregnant or lactating patients.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Clinical attachment level at 3 months in chronic periodontitis patients | 3 months
  The present randomized clinical trial assessed the effects of moxifloxacin, compared with chlorhexidine, locally administered via in situ gel formulation, on various clinical parameters describing periodontitis.

CONTACTS AND LOCATIONS:
Overall Officials: Shaurya Manjunath, MDS, Principal Investigator — Rajiv Gandhi University of Health Sceinces, Bangalore,Karnataka, India
Locations (1):
- Sri Hasanamba Dental College & Hospital, Hassan, Karnataka, India

REFERENCES:
- [Background] Guentsch A, Jentsch H, Pfister W, Hoffmann T, Eick S. Moxifloxacin as an adjunctive antibiotic in the treatment of severe chronic periodontitis. J Periodontol. 2008 Oct;79(10):1894-903. doi: 10.1902/jop.2008.070493. PMID 18834244